CLINICAL TRIAL: NCT05496322
Title: Continuous Vs Intermittent Non Invasive Blood Pressure Monitoring in Preventing Post Operative Organ Failure
Acronym: NiMon
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Collaborators: Societa Italiana Anestesia Analgesia Rianimazione e Terapia Intensiva (Other)
Responsible Party: Principal Investigator, Alberto Noto, Prof., University of Messina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-22
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure Determination; Hemodynamic Monitoring; Postoperative Complications
Keywords: Volume clamp; Continuous non invasive blood pressure monitoring
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- cNIBP (Experimental): Continuous non invasive blood pressure monitor (Volume clamp)
  Interventions: Device: Continuous Non Invasive Blood Pressure Monitoring
- iNIBP (Active Comparator): Intermittent Non Invasive Blood Pressure (Brachial Cuff)
  Interventions: Device: Intermittent Non Invasive Blood Pressure Monitoring

INTERVENTIONS:
Device: Continuous Non Invasive Blood Pressure Monitoring — Continuous non-invasive arterial pressure monitoring
  Arms: cNIBP
Device: Intermittent Non Invasive Blood Pressure Monitoring — Intermittent non-invasive arterial pressure monitoring
  Arms: iNIBP

SUMMARY:
Continuous non-invasive arterial pressure monitoring has the potential to decrease the duration of intraoperative hypotension and hypertension compared to conventional intermittent blood pressure monitoring. Chen et al. demonstrated using continuous non-invasive arterial pressure devices for every hour of surgery it is possible to identify an average of 14 minutes of potentially treatable hypotensive and hypertensive time(12). Whether the ability to detect more hypotension events by continuous non-invasive arterial pressure monitoring use can improve patient outcomes, is still an open research question

ELIGIBILITY:
Inclusion Criteria:

* All adult (age ≥18 years) patients scheduled for elective non-cardiac surgery in participating centers
* Surgical case planned with non invasive blood pressure monitoring according to local clinical practice or policies.

Exclusion Criteria:

* Missing of preoperative serum creatinine during 30 days prior surgery
* Preoperative dialysis
* Chronic kidney disease (eGFR < 60ml/min Cockcroft-Gault equation)
* Surgical procedure lasting less than 60 min
* Planned use of permissive hypotension
* Urological procedures (including nephrectomy and renal transplantation)
* Refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1265 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Post operative myocardial injury | 1 week
  The primary outcome will be the proportions of myocardial injury (Definitions: elevation of serum Troponin T (TnT) >= 30 ng/L in the first post-operative week)

SECONDARY OUTCOMES:
Post operative Acute kidney injury | 1 week
  Proportions of postoperative AKI (Definition: increase in postoperative serum creatinine concentration during the first 7 postoperative days by more than 1.5-fold or greater than 0.3 mg/dl. Preoperative concentration was defined as the most recent recorded measurement within 30 days before the surgery)
Post operative death | 28 day after surgery
  Death during postoperative hospital stay
Events 30d post surgery | 30 days after surgery
  Any of the following events after surgery: Stroke, Non fatal cardiac arrest, AKI stage 2-3, Sepsis, Death)
Events 90d post surgery | 90 days after surgery
  Any of the following events after surgery: Stroke, Non fatal cardiac arrest, AKI stage 2-3, Sepsis, Death)

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U. G.Martino - University of Messina, Messina, Italy

REFERENCES:
- [Derived] Noto A, Chalkias A, Madotto F, Ball L, Bignami EG, Cecconi M, Guarracino F, Messina A, Morelli A, Princi P, Sanfilippo F, Scolletta S, Tritapepe L, Cortegiani A; SIAARTI Study Group. Continuous vs intermittent Non-Invasive blood pressure MONitoring in preventing postoperative organ failure (niMON): study protocol for an open-label, multicenter randomized trial. J Anesth Analg Crit Care. 2024 Feb 6;4(1):7. doi: 10.1186/s44158-024-00142-w. PMID 38321507